CLINICAL TRIAL: NCT00474175
Title: Benzocaine Gel Toothache Dose-Response Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Collaborators: Church & Dwight Company, Inc. (Industry); Consumer Healthcare Products Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BZ-03-07; NCT00836511 (obsolete NCT alias)
Record Dates: First submitted 2007-05-14; First posted 2007-05-16 (Estimated); Results first posted 2012-01-18 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Toothache
MeSH Terms: conditions — Toothache | interventions — Benzocaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): Placebo control
  Interventions: Drug: Placebo gel
- 2 (Active Comparator): 10% benzocaine gel formulation
  Interventions: Drug: benzocaine
- 3 (Active Comparator): 20% benzocaine gel formulation
  Interventions: Drug: benzocaine

INTERVENTIONS:
Drug: Placebo gel — single dose (less than 1g) of a matching placebo gel
  Arms: 1
Drug: benzocaine — single dose (less than 1g) of 10% benzocaine gel formulation
  Arms: 2
Drug: benzocaine — single dose (less than 1g) of 20% benzocaine gel formulation
  Arms: 3

SUMMARY:
To evaluate the efficacy and safety of benzocaine gel products for the relief of toothache and to assess the subject's compliance with proposed label directions.

ELIGIBILITY:
Inclusion Criteria:

* Males or females at least 12 years of age.
* Presence of spontaneous toothache pain in only one permanent tooth. Toothache pain is due only to an open tooth cavity and only as a result of dental caries, loss of a restoration or tooth fracture.
* To qualify for the study, the subject must have a rating of at least moderate pain on the Dental Pain Scale (DPS) and a score of at least 50 mm on the Visual Analog Scale. To be included in the moderate pain stratum, the subjects must have a rating of moderate pain in the DPS and to be included in the severe pain stratum the subjects must have a rating of severe pain in the DPS.
* Females who are neither pregnant, as verified by a urine-based pregnancy test, nor breast-feeding.
* Female subjects of childbearing potential and those who are post-menopausal for less than 2 years must be using a medically approved method of contraception (i.e., oral, transdermal or implanted contraceptive devices, intrauterine device, diaphragm, condom, abstinence, or surgical sterility).
* Subjects must be reliable, cooperative and of adequate intelligence to read and understand the rating scales and other study instructions.
* Subjects must be able to read, comprehend, and sign the consent form. Minors will provide assent to study participation if age appropriate. Parent/legal guardian must be able to read, comprehend, and sign the informed consent form.

Exclusion Criteria:

* Presence of spontaneous toothache pain in a primary tooth. Presence of spontaneous toothache pain in more than one tooth. Presence of an open tooth cavity in a tooth adjacent to the painful tooth with the open tooth cavity.
* Presence of concomitant oral pain due to any other condition such as: soft-tissue lesions (e.g., aphthous or traumatic ulcer, herpes labialis, acute necrotizing ulcerative gingivitis); or multiple hard-tissue (e.g., carious) lesions; pain due to other surgical procedures, injuries or dental surface sensitivity.
* Presence of a periodontal abscess as diagnosed from an X-ray or clinical examination of the painful tooth.
* Presence of glucose-6-phosphate dehydrogenase (G6PD) deficiency.
* History of acute or chronic hemolytic anemia.
* History of sensitivity or allergy to benzocaine or other local anesthetic agents.
* Use of any short-acting oral or topical analgesic/ anesthetic product within 2 hours of enrollment or any long-acting Rx or OTC analgesic product within 4 hours of enrollment.
* Use of an investigational drug or participation in an investigational study within the past 30 days.
* Previous participation in this study.
* Member or a relative of the study site staff or sponsor directly involved in the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 577 (Actual)
Dates: Start 2007-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- United States (8):
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Buffalo, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=BZ-03-07&StudyName=Benzocaine%20Gel%20Toothache%20Dose-Response%20Study

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Single dose of placebo gel matched to either 10 % or 20 % benzocaine gel administered as per product label directions.
- Benzocaine 10%: Single dose of 10% benzocaine gel administered as per product label directions.
- Benzocaine 20%: Single dose of 20% benzocaine gel administered as per product label directions.
Period: Overall Study
Arm/Group | Placebo | Benzocaine 10% | Benzocaine 20%
Started | 115 | 233 | 229
Treated | 115 | 233 | 228
Completed | 114 | 226 | 225
Not Completed | 1 | 7 | 4
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Ineligible | 1 | 3 | 1
Not completed — Protocol Violation | 0 | 2 | 1
Not completed — Administrative | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Benzocaine 10% | Benzocaine 20% | Total
Number analyzed (Participants) | 115 | 233 | 228 | 576
Age Continuous [Mean (Standard Deviation); unit: Years] — Demographic data is only available for 576 participants who received study medication, except 1 participant who was randomized but not treated.
  Years | 31.2 (12.6) | 30.8 (12.7) | 31.3 (12.8) | 31.1 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Demographic data is only available for 576 participants who received study medication, except 1 participant who was randomized but not treated.
  Participants
    Female | 62 | 120 | 118 | 300
    Male | 53 | 113 | 110 | 276

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Response
Description: Responder was defined as participant experiencing improvement in pain intensity, as exhibited by a pain score reduction on the Dental Pain Scale (DPS) from baseline of at least 1 unit for two consecutive assessments anytime between the 5 and 20-minute time points. Response in DPS scale was assigned values as 0 (None), 1 (Mild), 2 (Moderate) and 3 (Severe).
Time Frame: Baseline, 5, 10, 15 and 20 minutes
Population: Intent to treat (ITT) population included all randomized participants who received study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Benzocaine 10% | Benzocaine 20%
Number analyzed (Participants) | 115 | 233 | 228
Percentage of participants | 70.4 | 80.7 | 87.3
Statistical Analysis 1: Comparison: Placebo vs Benzocaine 20%; P-value was calculated using Cochran-Mantel-Haenszel (CMH) test which was adjusted for site and baseline DPS. Treatment difference (Benzocaine 20% - Placebo) and its associated confidence interval (C.I.) was calculated based on CMH weighted percentages and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Alternative hypotheses tested in the study was that benzocaine 20% was significantly (p less than or equal to [=<] 0.05) more effective than placebo; Treatment difference = 16.46, 95% CI 2-sided [7.2 to 25.7]
Statistical Analysis 2: Comparison: Placebo vs Benzocaine 10%; P-value was calculated using CMH test which was adjusted for site and baseline DPS. Treatment difference (Benzocaine 10% - Placebo) and its associated C.I. was calculated based on CMH weighted percentages and the corresponding standard error; Test type: Superiority or Other; p = 0.038, Cochran-Mantel-Haenszel — Alternative hypotheses tested in the study was that benzocaine 10% was significantly (p=<0.05) more effective than placebo provided that benzocaine 20% was more effective than placebo; Treatment difference = 9.80, 95% CI 2-sided [0.3 to 19.3]
Statistical Analysis 3: Comparison: Benzocaine 10% vs Benzocaine 20%; P-value was calculated using CMH test which was adjusted for site and baseline DPS. Treatment difference (Benzocaine 20% - Benzocaine 10%) and its associated C.I. was calculated based on CMH weighted percentages and the corresponding standard error; Test type: Superiority or Other; p = 0.047, Cochran-Mantel-Haenszel; Dose response was considered established if the percentage of responders between the 20% and 10% was greater than or equal to 5%; Treatment difference = 6.72, 95% CI 2-sided [0.2 to 13.3]

2. Secondary Outcome: Time to First Confirmed Perceptible Relief
Description: Participants evaluated the time to first perceptible relief by stopping a stopwatch labeled 'first perceptible relief' at the moment they first began to experience any relief. Stopwatch was active up to 120 minutes after dosing or until stopped by the participant, or rescue medication was administered.
Time Frame: 0 to 120 minutes
Population: ITT population included all randomized participants who received study medication.
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Placebo | Benzocaine 10% | Benzocaine 20%
Number analyzed (Participants) | 115 | 233 | 228
Minutes | 2.0 [1.6 to 3.3] | 1.4 [1.2 to 1.7] | 1.1 [1.0 to 1.3]
Statistical Analysis 1: Comparison: Placebo vs Benzocaine 20%; P-value was calculated using Cox proportional hazard regression model which was adjusted for treatment, site and baseline DPS. Hazard Ratio (HR) of Benzocaine 20% relative to the Placebo was calculated. C.I. was based on the Wald statistic; Test type: Superiority or Other; p < 0.001, Regression, Cox — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Hazard Ratio (HR) = 2.02, 95% CI 2-sided [1.55 to 2.64]
Statistical Analysis 2: Comparison: Placebo vs Benzocaine 10%; P-value was calculated using Cox proportional hazard regression model which was adjusted for treatment, site and baseline DPS. HR of Benzocaine 10% relative to the Placebo was calculated. C.I. was based on the Wald statistic; Test type: Superiority or Other; p < 0.001, Regression, Cox — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Hazard Ratio (HR) = 1.63, 95% CI 2-sided [1.26 to 2.12]
Statistical Analysis 3: Comparison: Benzocaine 10% vs Benzocaine 20%; P-value was calculated using Cox proportional hazard regression model which was adjusted for treatment, site and baseline DPS. HR of Benzocaine 20% relative to the Benzocaine 10% was calculated. C.I. was based on the Wald statistic; Test type: Superiority or Other; p = 0.030, Regression, Cox — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Hazard Ratio (HR) = 1.24, 95% CI 2-sided [1.02 to 1.51]

3. Secondary Outcome: Time to Meaningful Relief
Description: Participants evaluated the time to meaningful relief by stopping a second stopwatch labeled 'meaningful relief' at the moment they first began to experience meaningful relief. Stopwatch was active up to 120 minutes after dosing or until stopped by the participant, or rescue medication was administered.
Time Frame: 0 to 120 minutes
Population: ITT population included all randomized participants who received study medication.
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Placebo | Benzocaine 10% | Benzocaine 20%
Number analyzed (Participants) | 115 | 233 | 228
Minutes | 8.5 [5.1 to 15.4] | 4.4 [3.7 to 5.8] | 3.2 [2.8 to 4.2]
Statistical Analysis 1: Comparison: Placebo vs Benzocaine 20%; P-value was calculated using Cox proportional hazard regression model which was adjusted for treatment, site and baseline DPS. HR of Benzocaine 20% relative to the Placebo was calculated. C.I. was based on the Wald statistic; Test type: Superiority or Other; p < 0.001, Regression, Cox — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Hazard Ratio (HR) = 2.04, 95% CI 2-sided [1.57 to 2.66]
Statistical Analysis 2: Comparison: Placebo vs Benzocaine 10%; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p < 0.001, Regression, Cox — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Hazard Ratio (HR) = 1.73, 95% CI 2-sided [1.34 to 2.25]
Statistical Analysis 3: Comparison: Benzocaine 10% vs Benzocaine 20%; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.100, Regression, Cox — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Hazard Ratio (HR) = 1.18, 95% CI 2-sided [0.97 to 1.43]

4. Secondary Outcome: Duration of Effect
Description: Duration of effect was defined as the time difference between onset of effect and its offset. Onset of effect was the first time point at which two consecutive pain scores less severe than at baseline by at least 1 unit (on the DPS) were attained. Offset of effect was the first of the following events to occur after onset: time to drop out if the drop out was due to lack of efficacy, time of rescue medication, or the first time point following onset of effect at which two consecutive pain scores that are at least as severe as at baseline were attained.
Time Frame: 0 to 120 minutes
Population: ITT population included all randomized participants who received study medication.
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Placebo | Benzocaine 10% | Benzocaine 20%
Number analyzed (Participants) | 115 | 233 | 228
Minutes | NA [NA to NA] — Data was not summarized as median time to duration of effect was greater than (>) 115 minutes for all treatment groups and therefore 95% C.I. was not estimable. | NA [NA to NA] — Data was not summarized as median time to duration of effect was >115 minutes for all treatment groups and therefore 95% C.I. was not estimable. | NA [NA to NA] — Data was not summarized as median time to duration of effect was >115 minutes for all treatment groups and therefore 95% C.I. was not estimable.

5. Secondary Outcome: Sum of Pain Relief Combined With Pain Intensity Differences (SPRID) Scores
Description: SPRID is time-weighted sum of pain relief scores combined with pain intensity difference (PRID) scores over 60 and 120 minutes. SPRID score range was 0 (worst) to 7 (best) for SPRID 60 and 0 (worst) to 14 (best) for SPRID 120. PRID is sum of Pain intensity differences (PID) and Dental pain relief scale (DPRS) scores at each post-dosing time point. PID was calculated as baseline DPS minus DPS score at given time point (DPS range: 0 [none] to 3 [severe]; baseline DPS range from 2-3). PID score ranges from -1 (worst) to 3 (best). DPRS is 5-point scale ranging from 0 (No-relief) to 4 (Complete).
Time Frame: 60 minutes and 120 minutes
Population: ITT population included all randomized participants who received study medication.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Benzocaine 10% | Benzocaine 20%
Number analyzed (Participants) | 115 | 233 | 228
Units on a scale
  SPRID 60 | 3.1 (2.3) | 3.4 (2.0) | 3.6 (2.0)
  SPRID 120 | 5.9 (4.8) | 6.4 (4.2) | 6.7 (4.3)
Statistical Analysis 1: Comparison: Placebo vs Benzocaine 20%; SPRID 60: P-value was calculated using Analysis of Variance (ANOVA) which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 20% - Placebo) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.035, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.49, 95% CI 2-sided [0.03 to 0.95]
Statistical Analysis 2: Comparison: Placebo vs Benzocaine 10%; SPRID 60: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 10% - Placebo) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.173, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.32, 95% CI 2-sided [-0.14 to 0.78]
Statistical Analysis 3: Comparison: Benzocaine 10% vs Benzocaine 20%; SPRID 60: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 20% - Benzocaine 10%) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.358, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.18, 95% CI 2-sided [-0.20 to 0.55]
Statistical Analysis 4: Comparison: Placebo vs Benzocaine 20%; SPRID 120: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 20% - Placebo) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.135, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.75, 95% CI 2-sided [-0.23 to 1.72]
Statistical Analysis 5: Comparison: Placebo vs Benzocaine 10%; SPRID 120: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 10% - Placebo) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.332, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.48, 95% CI 2-sided [-0.49 to 1.46]
Statistical Analysis 6: Comparison: Benzocaine 10% vs Benzocaine 20%; SPRID 120: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 20% - Benzocaine 10%) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.517, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.26, 95% CI 2-sided [-0.53 to 1.06]

6. Secondary Outcome: Time to Dropping Out Due to Lack of Efficacy or Rescue Medication
Description: Median time of dropping out of the participants from the study due to lack of efficacy or rescue medication (ibuprofen 200-400 mg or acetaminophen 1000 mg), whichever comes first.
Time Frame: 0 to 120 minutes
Population: ITT population included all randomized participants who received study medication.
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Placebo | Benzocaine 10% | Benzocaine 20%
Number analyzed (Participants) | 115 | 233 | 228
Minutes | NA [NA to NA] — Data was not summarized as median time for dropping out due to lack of efficacy or taking rescue medication for all treatment groups was >120 minutes (study duration) and therefore 95% C.I. was not estimable. | NA [NA to NA] — Data was not summarized as median time for dropping out due to lack of efficacy or taking rescue medication for all treatment groups was >120 minutes (study duration) and therefore 95% C.I. was not estimable. | NA [NA to NA] — Data was not summarized as median time for dropping out due to lack of efficacy or taking rescue medication for all treatment groups was >120 minutes (study duration) and therefore 95% C.I. was not estimable.

7. Secondary Outcome: Pain Relief Combined With Pain Intensity Difference (PRID) Scores
Description: PRID is sum of PID and DPRS scores at each post-dosing time point. The overall possible score range, for PRID is -1 (worst) to 7 (best). PID was calculated as baseline DPS minus DPS score at given time point (DPS range from 0 [none] to 3 [severe]; baseline DPS range from 2-3). PID score ranges from -1 (worst) to 3 (best). DPRS is 5-point scale ranging from 0 (No-relief) to 4 (Complete).
Time Frame: 5 to 120 minutes
Population: ITT population included all randomized participants who received study medication.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Benzocaine 10% | Benzocaine 20%
Number analyzed (Participants) | 115 | 233 | 228
Units on a scale
  5 minutes | 2.72 (2.05) | 3.25 (1.98) | 3.66 (1.87)
  10 minutes | 3.08 (2.25) | 3.56 (2.00) | 3.88 (1.97)
  15 minutes | 3.18 (2.46) | 3.64 (2.23) | 3.96 (2.07)
  20 minutes | 3.21 (2.50) | 3.64 (2.27) | 3.74 (2.23)
  25 minutes | 3.12 (2.53) | 3.60 (2.25) | 3.73 (2.27)
  30 minutes | 3.11 (2.65) | 3.39 (2.32) | 3.66 (2.38)
  40 minutes | 3.06 (2.60) | 3.44 (2.39) | 3.52 (2.43)
  50 minutes | 3.20 (2.68) | 3.41 (2.40) | 3.42 (2.45)
  60 minutes | 3.17 (2.74) | 3.18 (2.47) | 3.38 (2.57)
  70 minutes | 2.98 (2.75) | 3.16 (2.49) | 3.33 (2.59)
  80 minutes | 2.91 (2.77) | 3.09 (2.55) | 3.24 (2.60)
  90 minutes | 2.78 (2.70) | 3.05 (2.63) | 3.09 (2.61)
  100 minutes | 2.78 (2.70) | 3.00 (2.62) | 2.93 (2.58)
  110 minutes | 2.70 (2.71) | 2.90 (2.60) | 2.96 (2.59)
  120 minutes | 2.73 (2.72) | 2.82 (2.61) | 2.84 (2.56)
Statistical Analysis 1: Comparison: Placebo vs Benzocaine 20%; 5 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 20% - Placebo) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p < 0.001, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.93, 95% CI 2-sided [0.50 to 1.35]
Statistical Analysis 2: Comparison: Placebo vs Benzocaine 10%; 5 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 10% - Placebo) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.011, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.55, 95% CI 2-sided [0.13 to 0.97]
Statistical Analysis 3: Comparison: Benzocaine 10% vs Benzocaine 20%; 5 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 20% - Benzocaine 10%) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.031, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.38, 95% CI 2-sided [0.03 to 0.72]
Statistical Analysis 4: Comparison: Placebo vs Benzocaine 20%; 10 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 20% - Placebo) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p < 0.001, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.78, 95% CI 2-sided [0.33 to 1.23]
Statistical Analysis 5: Comparison: Placebo vs Benzocaine 10%; 10 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 10% - Placebo) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.031, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.49, 95% CI 2-sided [0.04 to 0.94]
Statistical Analysis 6: Comparison: Benzocaine 10% vs Benzocaine 20%; 10 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 20% - Benzocaine 10%) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.119, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.29, 95% CI 2-sided [-0.07 to 0.66]
Statistical Analysis 7: Comparison: Placebo vs Benzocaine 20%; 15 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 20% - Placebo) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.002, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.77, 95% CI 2-sided [0.28 to 1.25]
Statistical Analysis 8: Comparison: Placebo vs Benzocaine 10%; 15 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 10% - Placebo) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.061, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.46, 95% CI 2-sided [-0.02 to 0.95]
Statistical Analysis 9: Comparison: Benzocaine 10% vs Benzocaine 20%; 15 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 20% - Benzocaine 10%) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.131, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.30, 95% CI 2-sided [-0.09 to 0.70]
Statistical Analysis 10: Comparison: Placebo vs Benzocaine 20%; 20 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 20% - Placebo) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.044, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.52, 95% CI 2-sided [0.01 to 1.03]
Statistical Analysis 11: Comparison: Placebo vs Benzocaine 10%; 20 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 10% - Placebo) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.099, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.43, 95% CI 2-sided [-0.08 to 0.93]
Statistical Analysis 12: Comparison: Benzocaine 10% vs Benzocaine 20%; 20 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 20% - Benzocaine 10%) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.647, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.10, 95% CI 2-sided [-0.32 to 0.51]
Statistical Analysis 13: Comparison: Placebo vs Benzocaine 20%; 25 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 20% - Placebo) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.023, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.60, 95% CI 2-sided [0.08 to 1.11]
Statistical Analysis 14: Comparison: Placebo vs Benzocaine 10%; 25 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 10% - Placebo) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.072, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.47, 95% CI 2-sided [-0.04 to 0.98]
Statistical Analysis 15: Comparison: Benzocaine 10% vs Benzocaine 20%; 25 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 20% - Benzocaine 10%) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.551, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.13, 95% CI 2-sided [-0.29 to 0.55]
Statistical Analysis 16: Comparison: Placebo vs Benzocaine 20%; 30 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 20% - Placebo) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.047, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.54, 95% CI 2-sided [0.01 to 1.08]
Statistical Analysis 17: Comparison: Placebo vs Benzocaine 10%; 30 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 10% - Placebo) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.316, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.27, 95% CI 2-sided [-0.26 to 0.81]
Statistical Analysis 18: Comparison: Benzocaine 10% vs Benzocaine 20%; 30 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 20% - Benzocaine 10%) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.224, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.27, 95% CI 2-sided [-0.17 to 0.71]
Statistical Analysis 19: Comparison: Placebo vs Benzocaine 20%; 40 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 20% - Placebo) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.099, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.46, 95% CI 2-sided [-0.09 to 1.01]
Statistical Analysis 20: Comparison: Placebo vs Benzocaine 10%; 40 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 10% - Placebo) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.186, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.37, 95% CI 2-sided [-0.18 to 0.92]
Statistical Analysis 21: Comparison: Benzocaine 10% vs Benzocaine 20%; 40 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 20% - Benzocaine 10%) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.684, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.09, 95% CI 2-sided [-0.35 to 0.54]
Statistical Analysis 22: Comparison: Placebo vs Benzocaine 20%; 50 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 20% - Placebo) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.452, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.21, 95% CI 2-sided [-0.34 to 0.76]
Statistical Analysis 23: Comparison: Placebo vs Benzocaine 10%; 50 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 10% - Placebo) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.479, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.20, 95% CI 2-sided [-0.35 to 0.75]
Statistical Analysis 24: Comparison: Benzocaine 10% vs Benzocaine 20%; 50 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 20% - Benzocaine 10%) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.955, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.01, 95% CI 2-sided [-0.44 to 0.46]
Statistical Analysis 25: Comparison: Placebo vs Benzocaine 20%; 60 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 20% - Placebo) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.465, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.21, 95% CI 2-sided [-0.36 to 0.79]
Statistical Analysis 26: Comparison: Placebo vs Benzocaine 10%; 60 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 10% - Placebo) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.992, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.00, 95% CI 2-sided [-0.57 to 0.58]
Statistical Analysis 27: Comparison: Benzocaine 10% vs Benzocaine 20%; 60 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 20% - Benzocaine 10%) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.376, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.21, 95% CI 2-sided [-0.26 to 0.68]
Statistical Analysis 28: Comparison: Placebo vs Benzocaine 20%; 70 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 20% - Placebo) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.229, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.36, 95% CI 2-sided [-0.22 to 0.93]
Statistical Analysis 29: Comparison: Placebo vs Benzocaine 10%; 70 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 10% - Placebo) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.581, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.16, 95% CI 2-sided [-0.41 to 0.74]
Statistical Analysis 30: Comparison: Benzocaine 10% vs Benzocaine 20%; 70 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 20% - Benzocaine 10%) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.422, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.19, 95% CI 2-sided [-0.28 to 0.66]
Statistical Analysis 31: Comparison: Placebo vs Benzocaine 20%; 80 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 20% - Placebo) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.271, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.33, 95% CI 2-sided [-0.26 to 0.91]
Statistical Analysis 32: Comparison: Placebo vs Benzocaine 10%; 80 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 10% - Placebo) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.612, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.15, 95% CI 2-sided [-0.43 to 0.73]
Statistical Analysis 33: Comparison: Benzocaine 10% vs Benzocaine 20%; 80 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 20% - Benzocaine 10%) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.465, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.18, 95% CI 2-sided [-0.30 to 0.65]
Statistical Analysis 34: Comparison: Placebo vs Benzocaine 20%; 90 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 20% - Placebo) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.290, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.32, 95% CI 2-sided [-0.27 to 0.91]
Statistical Analysis 35: Comparison: Placebo vs Benzocaine 10%; 90 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 10% - Placebo) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.412, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.25, 95% CI 2-sided [-0.34 to 0.83]
Statistical Analysis 36: Comparison: Benzocaine 10% vs Benzocaine 20%; 90 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 20% - Benzocaine 10%) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.769, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.07, 95% CI 2-sided [-0.41 to 0.55]
Statistical Analysis 37: Comparison: Placebo vs Benzocaine 20%; 100 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 20% - Placebo) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.610, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.15, 95% CI 2-sided [-0.43 to 0.74]
Statistical Analysis 38: Comparison: Placebo vs Benzocaine 10%; 100 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 10% - Placebo) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.511, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.20, 95% CI 2-sided [-0.39 to 0.78]
Statistical Analysis 39: Comparison: Benzocaine 10% vs Benzocaine 20%; 100 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 20% - Benzocaine 10%) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.859, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = -0.04, 95% CI 2-sided [-0.52 to 0.43]
Statistical Analysis 40: Comparison: Placebo vs Benzocaine 20%; 110 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 20% - Placebo) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.386, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.26, 95% CI 2-sided [-0.33 to 0.84]
Statistical Analysis 41: Comparison: Placebo vs Benzocaine 10%; 110 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 10% - Placebo) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.563, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.17, 95% CI 2-sided [-0.41 to 0.76]
Statistical Analysis 42: Comparison: Benzocaine 10% vs Benzocaine 20%; 110 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 20% - Benzocaine 10%) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.721, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.09, 95% CI 2-sided [-0.39 to 0.56]
Statistical Analysis 43: Comparison: Placebo vs Benzocaine 20%; 120 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 20% - Placebo) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.725, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.10, 95% CI 2-sided [-0.48 to 0.69]
Statistical Analysis 44: Comparison: Placebo vs Benzocaine 10%; 120 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 10% - Placebo) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.839, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.06, 95% CI 2-sided [-0.52 to 0.64]
Statistical Analysis 45: Comparison: Benzocaine 10% vs Benzocaine 20%; 120 minutes: P-value was calculated using ANOVA which was adjusted for treatment, site and baseline DPS. Treatment difference (Benzocaine 20% - Benzocaine 10%) and corresponding 95% C.I. were calculated based on least-squares means from the ANOVA model with treatment, site, and baseline DPS effects; Test type: Superiority or Other; p = 0.855, ANOVA — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.04, 95% CI 2-sided [-0.43 to 0.52]

8. Secondary Outcome: Global Satisfaction Assessment
Description: Participants were asked to provide an overall assessment of their satisfaction with the study medication on a categorical scale. Response in this scale was assigned values as 0 (Poor), 1 (Fair), 2 (Good), 3 (Very Good) and 4 (Excellent).
Time Frame: 120 minutes
Population: ITT population included all randomized participants who received study medication.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Benzocaine 10% | Benzocaine 20%
Number analyzed (Participants) | 115 | 233 | 228
Units on a scale | 2.1 (1.6) | 2.5 (1.2) | 2.5 (1.2)
Statistical Analysis 1: Comparison: Placebo vs Benzocaine 20%; P-value was calculated from the CMH test with modified ridit scores, adjusted for site baseline pain intensity. Treatment difference (Benzocaine 20% versus Placebo) and the associated confidence interval were calculated based on the weighted Gamma statistic; Test type: Superiority or Other; p = 0.035, Cochran-Mantel-Haenszel — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.17, 95% CI 2-sided [0.01 to 0.33]
Statistical Analysis 2: Comparison: Placebo vs Benzocaine 10%; P-value was calculated from the CMH test with modified ridit scores, adjusted for site baseline pain intensity. Treatment difference (Benzocaine 10% versus Placebo) and the associated confidence interval were calculated based on the weighted Gamma statistic; Test type: Superiority or Other; p = 0.039, Cochran-Mantel-Haenszel — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = 0.16, 95% CI 2-sided [-0.00 to 0.33]
Statistical Analysis 3: Comparison: Benzocaine 10% vs Benzocaine 20%; P-value was calculated from the CMH test with modified ridit scores, adjusted for site baseline pain intensity. Treatment difference (Benzocaine 20% versus Benzocaine 10%) and the associated confidence interval were calculated based on the weighted Gamma statistic; Test type: Superiority or Other; p = 0.944, Cochran-Mantel-Haenszel — The a priori threshold p-value was specified as 0.05, and no adjustments were made for multiple comparisons; Treatment difference = -0.01, 95% CI 2-sided [-0.15 to 0.13]

9. Other Pre Specified Outcome: Dosing Compliance Calculated by Evaluating Amount of Study Medication Applied
Description: Amount of study medication applied was calculated by weighing medication tube prior and post-dosing.
Time Frame: Baseline and 5 minutes
Population: Safety population included all participants who received at least 1 dose of study medication and had follow up data.
Measure: Mean (Standard Deviation); unit: Milligram (mg)
Arm/Group | Placebo | Benzocaine 10% | Benzocaine 20%
Number analyzed (Participants) | 115 | 233 | 228
Milligram (mg) | 258.6 (163.4) | 226.8 (138.2) | 233.1 (150.7)

10. Other Pre Specified Outcome: Dosing Compliance Calculated by Evaluating Percentage of Participants Who Applied no More Than 400 mg of the Study Medication
Time Frame: Baseline and 5 minutes
Population: Safety population included all participants who received at least 1 dose of study medication and had follow up data.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Benzocaine 10% | Benzocaine 20%
Number analyzed (Participants) | 115 | 233 | 228
Percentage of participants | 83.5 [75.6 to 89.2] | 89.3 [84.6 to 92.6] | 89.5 [84.8 to 92.8]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo | Benzocaine 10% | Benzocaine 20%
Serious Adverse Events (participants affected / at risk) | 0/115 | 0/233 | 0/228
Other Adverse Events (participants affected / at risk) | 4/115 | 6/233 | 6/228
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=115) | Benzocaine 10% (N=233) | Benzocaine 20% (N=228)
Diplopia (Eye disorders) | 0 | 1 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 1
Stomach upset (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Post operation wound infection (Infections and infestations) | 1 | 0 | 0
Tooth caries Not Otherwise Specified (NOS) (Infections and infestations) | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 2 | 1
Somnolence (Nervous system disorders) | 1 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Nervousness (Psychiatric disorders) | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Wyeth has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.